CLINICAL TRIAL: NCT02018094
Title: A Randomised Control Trial to Determine Whether a 5 Day Course of Antibiotics is More Clinically and Cost Effective Than a 24 Hour Prophylactic Course for the Prevention of Surgical Site Infection Following Lower Limb Amputation
Brief Title: The Amputation Surgical Site Infection Trial (ASSIT)
Acronym: ASSIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ASSIT Trial
Record Dates: First submitted 2013-12-05; First posted 2013-12-23 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Wound Infection; Amputation Wound
Keywords: Amputation; Infection; Skin Preparation; SSI; Stump; Wound
MeSH Terms: conditions — Wound Infection; Infections; Wounds and Injuries | interventions — Amoxicillin-Potassium Clavulanate Combination; Iodine; Povidone-Iodine; Metronidazole; Chlorhexidine; Hydrex; Teicoplanin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 24 hour antibiotic course (Active Comparator): 24 hours of the stated antibiotics administered intravenously (Augmentin and metronidazole. Teicoplanin and or gentamicin will be used if penicillin allergic and state of renal function)
  Interventions: Drug: Co-amoxiclav; Drug: Iodine; Drug: Metronidazole; Drug: Chlorhexidine; Drug: Teicoplanin
- 5 day antibiotic Course (Active Comparator): 24 hours of IV antibiotics followed by 4 days of oral antibiotics (Augmentin and metronidazole. Teicoplanin and or gentamicin will be used if penicillin allergic and state of renal function. Clindamycin will be used as a an oral replacement for penicillin allergic patients)
  Interventions: Drug: Co-amoxiclav; Drug: Iodine; Drug: Metronidazole; Drug: Chlorhexidine; Drug: Teicoplanin; Drug: Clindamycin
- Iodine (Active Comparator): Skin Preparation used pre-operatively: Alcoholic Povidone
  Interventions: Drug: Co-amoxiclav; Drug: Iodine; Drug: Metronidazole; Drug: Teicoplanin; Drug: Clindamycin
- Chlorhexidine (Active Comparator): Skin preparation to be used preoperatively: Alcoholic chlorhexidine
  Interventions: Drug: Co-amoxiclav; Drug: Metronidazole; Drug: Chlorhexidine; Drug: Teicoplanin; Drug: Clindamycin

INTERVENTIONS:
Drug: Co-amoxiclav — Augmentin 1.2g IV three times daily for 24 hours. If the patient is randomised to the 5-day duration antibiotic arm then Augmentin 625mg oral tablets three times daily are added to the 24 hour course for a further 4 days.
  Other Names: Augmentin
Drug: Iodine — Intra-operative skin preparation prior to incision to skin.
  Other Names: Povidone iodine (alcoholic solution)
  Arms: 24 hour antibiotic course; 5 day antibiotic Course; Iodine
Drug: Metronidazole — 500mg IV three times daily for 24 hours. If the patient is randomised to 5-day duration arm, then another 4 days of oral metronidazole at 400mg three times daily is added to the course
  Other Names: Flagyl
Drug: Chlorhexidine — Alcoholic Chlorhexidine skin pre-op preparation
  Other Names: Hydrex
  Arms: 24 hour antibiotic course; 5 day antibiotic Course; Chlorhexidine
Drug: Teicoplanin — Teicoplanin 400mg on induction. If penicillin allergic and on 5-day antibiotic arm then add clindamycin 300mg 4 times daily for further 4 days
Drug: Clindamycin — Clindamycin 300mg 4 times daily orally to be used in case of penicillin allergy
  Arms: 5 day antibiotic Course; Chlorhexidine; Iodine

SUMMARY:
* Lower limb amputations are performed usually as a last resort in patients with acute and chronic limb ischaemia (CLI) caused by vascular disease, poorly controlled diabetes or, infection.
* In the period 2003-2008 there were approximately 5,000 amputations per year in the UK.
* The Centre for Disease Control defines a Surgical Site Infection (SSI) as an infection within 30 days of an operation or up to one year if an implant is left in place and the infection is related to an operative procedure.
* Figures from the Surgical Site Infection Surveillance reported that the highest rate of surgical site infection was reported in association with lower limb amputation at 13.1%.
* There is a clear under-representation and the infection rate within our institution is approximately 25% which reflects the infection rate reported in a recent trial by Sadat et al (22.5%)
* Prevention of surgical site infections is of paramount importance to patients, healthcare providers and policy-makers, as they impact on morbidity and mortality and have significant time and cost implications.
* Currently there is NO CONSENSUS as to what the best practice is towards antibiotic administration in such patients. From a questionnaire-based audit we performed including vascular departments across the entire country, practice varies in both course duration (single dose → 5 days antibiotic course) as well as choice of antibiotics.
* The guideline at our institution suggests the 5-day course of antibiotic prophylaxis. The course duration varies depending on the clinical picture as well as microbiology results and recommendations.
* There are no randomised control trials that have investigated this aspect of patient care. We have set up one such trial and through it, we are looking to establish a standard practice which will hopefully be as beneficial as possible to the patient but also cost-effective for NHS.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 yrs undergoing lower limb amputations who are able to consent to the trial.
2. Able to understand the Patient Information Sheet and capable and willing to give informed consent and follow the protocol requirements (including attending all follow-up visits)

Exclusion Criteria:

1. Allergies to chlorhexidine/ alcohol/ iodophors
2. Inability to give informed consent
3. Patients who are admitted to hospital with severe sepsis secondary to gas gangrene requiring multiple operations and admission to Intensive Care Unit.
4. Aged under 18 years at the time of recruitment
5. Use of investigational drug/device therapy within preceding 4 weeks that may interfere with this study.
6. Toe amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days
  Primary objective: to establish the effect of 5 days of antibiotics versus a 24-hour prophylactic course on the incidence of surgical site infection (SSI) - total ASEPSIS score >21

SECONDARY OUTCOMES:
Impact of different skin preparations on infection rates | 30 days
  ASEPSIS Questionnaire score >21
Rate of re-intervention | 30 days
  Types of re-intervention: angioplasty, bypass, debridement, revision to higher level amputation.
Mortality | 1 year
  Mortality of a patient
Satisfactory healing rates | 3 months
  Metric Measurement. Asepsis score derived by HPA post-discharge questionnaire. Clinical examination, quality of life, time to prosthesis also recorded.
Quality of life Questionnaire | 1 year
  Assessed with Short form (SF)-12 questionnaire
Resource use | up to 3 months
  length of stay, return to surgery, number of visits to general practitioners, hospital visits, and prescription of antibiotics.
Rate of C. Diff., MSSA (Methicillin Sensitive Staphylococcus Aureus), MRSA (Methicillin Resistant Staphylococcus Aureus) infection | 30 days
  Infection progress
Mobility | 1 year
  Locomotor Capabilities index - 5
Pain Control | 1 year
  McGill Pain questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom

REFERENCES:
- [Derived] Souroullas P, Barnes R, Carradice D, Smith G, Huang C, Chetter I. Extended-course antibiotic prophylaxis in lower limb amputation: randomized clinical trial. Br J Surg. 2022 Apr 19;109(5):426-432. doi: 10.1093/bjs/znac053. PMID 35325055